CLINICAL TRIAL: NCT06811610
Title: Reliability of a Portable Audiometric Device Based on Active Noise-Canceling Headphones for Clinical Hearing Assessment
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Collaborators: Wuhan Douting Technology Co., Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: KY20242145zhadingjun
Record Dates: First submitted 2025-01-22; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-03

CONDITIONS: Hearing Loss, Bilateral or Unilateral
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Gender, age, disease and threshold values for each frequency of both audiometry for each participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Participants were tested for hearing using a new type of hearing detection device — Participants' hearing was tested using a portable audiometry device (E200) based on active noise-cancelling headphones, manufactured by Wuhan Doulisten Technology Co., LTD
Diagnostic Test: Participants' hearing was tested using a new portable pure tone audiometry device — Participants' hearing was tested using a portable audiometry device (E200) based on active noise-cancelling headphones, manufactured by Wuhan Doulisten Technology Co., LTD

SUMMARY:
Part One: Research Background Globally, approximately 500 million people suffer from disabling hearing loss, accounting for about 6.8% of the world's population. Hearing loss has emerged as a major global health issue. The cornerstone of hearing loss prevention and protection lies in hearing level testing. Early detection and intervention are crucial components of hearing healthcare. Currently, pure tone audiometry serves as the gold standard for hearing level testing, requiring patients to visit a hospital's standard soundproof room and complete the test under the guidance of a professional audiologist. However, existing professional audiometers are bulky, consume high power, and necessitate soundproof rooms (with background noise <30dBA), among other drawbacks. Moreover, primary hospitals or units lack professional audiologists and soundproof rooms, making it impossible to diagnose and treat hearing loss. Therefore, a portable hearing testing device that does not require a soundproof room would be a boon for the diagnosis and treatment of hearing loss patients. Currently, Wuhan Douting Technology Co., Ltd. has produced a portable hearing testing device (E200), supporting frequencies from 125Hz to 16000Hz, covering both conventional and extended high frequencies. The frequency tolerance, total harmonic distortion, and accuracy of hearing levels fully meet the technical requirements of Grade 4 audiometers according to national standards. In addition to meeting the functional and performance requirements of general audiometers, this device offers the following technical advantages and innovations: 1. Combining active and passive noise reduction, it achieves comprehensive noise reduction of over 29dBSPL, allowing for audiometry in environments with background noise <60dBA; 2. Supporting extended high frequencies, it can detect potential hearing damage earlier; 3. Supporting audiometry for rapid use by non-professionals, with automatic calibration, allowing non-professionals to operate by following prompts. This device is not yet on the market, and we intend to verify its reliability in assessing hearing conditions.

Part Two: Research Objectives To verify the reliability of a novel portable hearing testing device in assessing hearing conditions.

Part Three: Research Design Paired design

Part Four: Inclusion and Exclusion Criteria

Inclusion Criteria:

Age: ≥6 years old, no gender restriction Able to cooperate in completing pure tone audiometry

Exclusion Criteria:

Patients with acute otitis media or unremovable secretions blocking the external auditory canal Patients with mental or psychological disorders or unable to cooperate with the examination for other reasons

Part Five: Research Process This study will recruit volunteers from the outpatient and inpatient departments of Xijing Hospital. Each volunteer will undergo two audiological tests, with at least a 10-minute interval between the two tests to prevent intolerance to the hearing tests. Each audiological test will take approximately 6-8 minutes per subject.

Consultation and Physical Examination:

Researchers will collect general information, including name, gender, age, hearing status, and ear disease history; Conduct a physical examination of the ears; If a volunteer meets the inclusion criteria and voluntarily sign the informed consent form, researchers will determine the testing order using a random number method based on your enrollment sequence.

Conventional pure-tone audiometry:Patients undergo conventional pure tone audiometry using the interacoustics AC40 (Denmark) with TDH39 headphones (Telephonics; Farmingdale, NY, USA). We conducte audiometric testing in a sound-proof booth (background noise<30dBA) and evaluate the frequency range of 125-8000 Hz. Before the audiometry, patients will be asked to identify which ear have better hearing, and the ear with better hearing was tested first. This study employ the Hughson-Westlake approach, known as the " up-5 down-10 technique." The pure tone sound level was initially introduced at an estimated higher threshold and reduced by 10 dB HL after a correct response from the patient. If the patient did not respond correctly or at all, the sound level was increased by 5 dB HL. When there was a difference of 40 dB HL or more in air conduction thresholds between the ears, contralateral masking was applied to correct the cross-hearing.

E200 Audiometry: Noise-canceling headphones (RAN-3500) are used for all patients during the E200 audiometry. This is conducted in a regular room (ambient noise: 42.6-58.7 dBA, measured using a standard sound level meter: AWA6292 Multi-function Sound Level Meter) adjacent to a busy hallway without a sound-proof booth to simulate an ordinary environment. The Hughson-Westlake approach and contralateral masking are applied when conducting the E200 audiometry.

DETAILED DESCRIPTION:
Quality Control： Double-blind: The examiner does not have access to the results of the other testing technique until the experiment is completed, and the patient remains unaware of the results of both testing approaches until the end of the experiment.

Randomization: The sequence in which the patient undergoes the hearing tests is randomly determined using a random number table, ensuring an interval of at least 10 min between the two tests to avoid errors caused by fatigue or discomfort from consecutive testing.

Two individuals were responsible for entering the data, after which they verified each other's entries for accuracy.

Risks and Discomforts:

This study is a paired study utilizing a crossover trial method. All participants will undergo non-invasive procedures including basic information collection, medical history inquiry, physical examination, and pure tone audiometry. Pure tone audiometry, a standard outpatient clinical test, is conducted in a soundproof room. While this is a commonly used clinical examination method, an extremely small number of subjects may experience discomfort such as nervousness and anxiety due to不适应 to the enclosed environment. These symptoms can quickly subside once the subject leaves the environment and generally do not require special treatment. During the hearing test, pure tones are used. A minority of subjects with acoustic sensitivity may experience intolerance, ear pain, or other discomfort when exposed to louder sound stimuli. To mitigate this, the sound is gradually increased from a low volume during the examination. The researcher will closely monitor the subject's reactions, and if discomfort arises, the examination will be immediately halted. In most cases, symptoms will spontaneously resolve without special treatment after the examination is stopped. This study does not pose any additional risks to participants. For any adverse reactions that occur during the study, the researcher must accurately record them, promptly handle them according to medical protocols, and increase the frequency of follow-up visits or conduct additional laboratory tests based on the subject's condition. Follow-up should continue until the issue is properly resolved, the subject's condition stabilizes or returns to normal, or the researcher deems it appropriate to terminate follow-up.

Personal Information Confidentiality:

The information collected in this study will be kept confidential within the hospital as confidential material. To protect the identity of the subjects, any information related to the subjects in the research documents will be identified using a uniformly formatted number rather than names. Among all the collected and combined information of the subjects, any information that could help identify you will be removed to ensure that the relevant information cannot be linked to a specific research subject.

Sample Size Calculation： Based on the 69 data groups obtained in the pre-experiment, the Kappa coefficients were calculated as follows: left ear: 0.764, right ear: 0.743. A confidence level of 0.9 (α= 0.1) was used, and the confidence interval width was set to 0.2. The sample sizes computed using the PASS 2021 were determined to be 89 for the left ear and 107 for the right ear (eFigure 2 in Supplement 1). Ultimately, 114 patients were enrolled to validate the reliability of the E200.

Ethics： All patients provided written informed consent, and the study was approved by the Medical Ethics Committee of the First Affiliated Hospital of the Air Force Medical University(Ethics Committee FILE No: KY20242145-F-1). This study was conducted in accordance with the Declaration of Helsinki and Good Clinical Practice guidelines .

ELIGIBILITY:
Inclusion Criteria:

* Age:≥6 years old, regardless of gender
* Must be able to cooperate in completing pure tone audiometry

Exclusion Criteria:

* Acute phase of otitis media or external ear canal within the secretion blockage can not be removed
* Those suffering from mental illness or other reasons unable to cooperate with the completion of the examination Remarks: Each participant was examined by a specialist using otoscope. Those with ceruminous external auditory canal embolism or secretion blockage were cleared before audiological examination

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Volunteers who need hearing testing (pure tone audiometry) for various reasons or diseases are recruited from the ENT outpatient clinic or ward of Xijing Hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Hearing thresholds of each frequency of two hearing detection methods | 2024.03.29-2026.06.30
  Each participant used standard soundproof room pure tone audiometry (gold standard) and a new portable audiometry. The hearing thresholds of each frequency obtained by the two methods were recorded for each volunteer and compared

CONTACTS AND LOCATIONS:
Overall Officials: dingjun zha, Doctor of Medicine, Study Director — Department of Otolaryngology, the First Affiliated Hospital of Air Force Medical University
Locations (1):
- The First Affiliated Hospital of the Air Force Medical University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes
all data can be provided except for personal information of the volunteer
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2026.03-2028.12
Access Criteria: All researchers who are interested in this study can obtain the original data of this study (excluding the personal information of volunteers, such as name, gender, age, disease, etc.). The available data include the hearing test results of each volunteer with two kinds of tests, the overall gender, age, and disease distribution of all volunteers, etc. They can obtain IPD by emailing the researcher at kydgao123@qq.com

REFERENCES:
- [Background] Lee SY, Seo HW, Jung SM, Lee SH, Chung JH. Assessing the accuracy and reliability of application-based audiometry for hearing evaluation. Sci Rep. 2024 Mar 28;14(1):7359. doi: 10.1038/s41598-024-57944-9. PMID 38548854